CLINICAL TRIAL: NCT00806845
Title: Gewinnung Humaner antikörperproduzierender Zellen Aus Dem Blut
Brief Title: Examination of B Cell Responses in Human Blood
Status: Completed | Type: Observational
Sponsor: Regenerative Medicine Network (Network)
Collaborators: University of Leipzig (Other)
Responsible Party: Principal Investigator, Christian Jassoy, Professor of Virology, Regenerative Medicine Network
Other Study IDs: RegMedNet-001
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections
Keywords: HIV; B-lymphocyte
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- HIV infected individuals, HIV controllers: CD4+ T cell count > 350/µl, HIV load < 1000 copies/ml
- HIV infected individuals, early progressors: CD4+ T cell count > 350/µl, HIV load > 1000 copies/ml
- HIV infected individuals, late progressors: CD4+ T cell count < 200/µl
- HIV infected individuals, late progressors with therapy: CD4+ T cell count < 200/µl, under ART
- Healthy individuals: Uninfected

SUMMARY:
The aim of this study is the assessment B-cell immune responses in HIV-infected individuals.

DETAILED DESCRIPTION:
Groups of patients with different immune competencies will be examined. The impact of HIV infection on immune response will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals
* controls

Exclusion Criteria:

- none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV patients and controls attending specialised clinics, Germany
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Antigen specific B-cell responses | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Jassoy, MD, Study Director — Universität Leipzig
Locations (1):
- Universität Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- [Result] Bussmann BM, Reiche S, Bieniek B, Krznaric I, Ackermann F, Jassoy C. Loss of HIV-specific memory B-cells as a potential mechanism for the dysfunction of the humoral immune response against HIV. Virology. 2010 Feb 5;397(1):7-13. doi: 10.1016/j.virol.2009.11.003. Epub 2009 Dec 4. PMID 19962720
- [Result] Kunz K, Reiche S, Dwai Y, Cordes C, Krznaric I, Bussmann BM, Jassoy C. A broad spectrum of functional HIV-specific memory B cells in the blood of infected individuals with high CD4+ T-cell counts. J Acquir Immune Defic Syndr. 2011 Jul 1;57(3):e56-8. doi: 10.1097/QAI.0b013e31821dd9d1. No abstract available. PMID 21860350
- [Result] Reiche S, Nestler C, Sieg M, Schulz K, Cordes C, Krznaric I, Jassoy C. Hepatitis C virus (HCV)-specific memory B-cell responses in transiently and chronically infected HIV positive individuals. J Clin Virol. 2014 Apr;59(4):218-22. doi: 10.1016/j.jcv.2014.01.023. Epub 2014 Feb 4. PMID 24566009